CLINICAL TRIAL: NCT00795145
Title: Single Dose Safety, Tolerability And Pharmacokinetics Of Escalating Intravenous Doses Of Linezolid Followed By Evaluation Of The Effect Of Single Intravenous Doses Of Linezolid On QTc Interval In Healthy Subjects
Brief Title: A Study To Assess The Effect Of Linezolid On QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A5951151
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-05

CONDITIONS: Bacterial Infections
Keywords: Linezolid, QTc interval, pharmacokinetics, therapeutic dose, supra-therapeutic dose
MeSH Terms: conditions — Bacterial Infections | interventions — Linezolid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 1: 900 mg linezolid (Experimental)
  Interventions: Drug: Linezolid 900 mg
- Cohort 1: 1200 mg linezolid (Experimental)
  Interventions: Drug: Linezolid 1200 mg
- Cohort 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2: 600 mg linezolid (Experimental)
  Interventions: Drug: Linezolid 600 mg
- Cohort 2: 1200 mg linezolid (Experimental)
  Interventions: Drug: Linezolid 1200 mg
- Cohort 2: 400 mg Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Placebo — Intravenous, Placebo control for blinding, Normal Saline, Single dose
  Arms: Cohort 1: Placebo
Drug: Linezolid 900 mg — Intravenous, 900 mg linezolid, single dose
  Other Names: Zyvox
  Arms: Cohort 1: 900 mg linezolid
Drug: Linezolid 1200 mg — Intravenous, 1200 mg linezolid, single dose
  Other Names: Zyvox
  Arms: Cohort 1: 1200 mg linezolid
Drug: Placebo — Intravenous, Placebo control for blinding, Normal Saline, Single dose
  Arms: Cohort 2: Placebo
Drug: Linezolid 600 mg — Intravenous, 600 mg linezolid, single dose
  Other Names: Zyvox
  Arms: Cohort 2: 600 mg linezolid
Drug: Linezolid 1200 mg — Intravenous, 1200 mg linezolid, single dose
  Other Names: Zyvox
  Arms: Cohort 2: 1200 mg linezolid
Drug: Moxifloxacin 400 mg — Oral, 400 mg moxifloxacin, single dose
  Other Names: Avelox
  Arms: Cohort 2: 400 mg Moxifloxacin

SUMMARY:
The FDA has asked Pfizer to assess the risk of linezolid on QT interval (obtained from ECG readings) which could predispose patients to ventricular arrhythmias. This study is conducted to satisfy this requirement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 21 and 55 years.
* Body mass Index (BMI) of 18 to 30 kg/m2; and a total body weight > 45 kg (99 lbs).
* An informed consent document signed and dated.

Exclusion Criteria:

* Evidence or history of clinically significant abnormality.
* 12-lead ECG demonstrating QTc >450 msec at Screening.
* Receiving selective serotonin reuptake inhibitors (SSRIs) and/or sympathomimetic agents.
* Abnormal liver function tests.
* A positive urine drug screen, history of excessive alcohol and tobacco use.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951151&StudyName=A%20Study%20To%20Assess%20The%20Effect%20Of%20Linezolid%20On%20QTc%20Interval

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Sequence 1: Subjects were randomly assigned to placebo first, then linezolid 900 milligrams (mg) followed by 1200 mg linezolid, after a washout period of 48 hours between doses in Sequence 1.
- Cohort 1: Sequence 2: Subjects were randomly assigned to linezolid 900 mg first, then placebo, followed by 1200 mg linezolid, after a washout period of 48 hours between doses in Sequence 2.
- Cohort 1: Sequence 3: Subjects were randomly assigned to linezolid 900 mg first, then 1200 mg linezolid, followed by placebo after a washout period of 48 hours between doses in Sequence 3.
- Cohort 2: Sequence 1: Subjects were randomly assigned to placebo, then moxifloxacin, followed by linezolid 600 mg and 1200 mg, after a washout period of 48 hours between doses in Sequence 1.
- Cohort 2: Sequence 2: Subjects were randomly assigned to linezolid 600 mg first, then linezolid 1200 mg followed by placebo and moxifloxacin, after a washout period of 48 hours between doses in Sequence 2.
- Cohort 2: Sequence 3: Subjects were randomly assigned to linezolid 1200 mg first, then moxifloxacin 400 mg followed by linezolid 600 mg and placebo after a washout period of 48 hours between doses in Sequence 3.
- Cohort 2: Sequence 4: Subjects were randomly assigned to moxifloxacin 400 mg first, then placebo followed by linezolid 1200 mg and 600 mg linezolid after a washout period of 48 hours between doses in Sequence 4.
Period: Cohort 1
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4
Started | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2
Arm/Group | Cohort 1: Sequence 1 | Cohort 1: Sequence 2 | Cohort 1: Sequence 3 | Cohort 2: Sequence 1 | Cohort 2: Sequence 2 | Cohort 2: Sequence 3 | Cohort 2: Sequence 4
Started | 0 | 0 | 0 | 10 | 10 | 10 | 10
Completed | 0 | 0 | 0 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Placebo, Linezolid 900 mg and 1200 mg: Subjects were randomly assigned to placebo followed by linezolid 900 mg then 1200 mg linezolid in Sequence 1; or, linezolid 900 mg then linezolid 1200 mg followed by placebo in Sequence 2; or, linezolid 900 mg then placebo followed by linezolid 1200 mg in Sequence 3. There was a washout period of 48 hours between doses.
- Cohort 2: Placebo, Linezolid 600 mg and 1200 mg, Moxifloxacin: Subjects were randomly assigned to placebo first then moxifloxacin followed by linezolid 600 mg and 1200 mg linezolid last in Sequence 1; or linezolid 600 mg first then linezolid 1200 mg followed by placebo and moxifloxacin last in Sequence 2; or, linezolid 1200 mg first then moxifloxacin 400 mg followed by linezolid 600 mg and placebo last in Sequence 3; or, moxifloxacin 400 mg first then placebo followed by linezolid 1200 mg and 600 mg linezolid last in Sequence 4. There was a washout period of 48 hours between each dose.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo, Linezolid 900 mg and 1200 mg | Cohort 2: Placebo, Linezolid 600 mg and 1200 mg, Moxifloxacin | Total
Number analyzed (Participants) | 9 | 40 | 49
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  18 - 44 years | 8 | 36 | 44
  45 - 64 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 20 | 24
  Male | 5 | 20 | 25

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product(s) were reported.
Time Frame: From the time the subject had taken at least one dose of study treatment up to 5 weeks
Population: Safety Analysis Set (SAS): All subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Cohort 1: Placebo: 600 milliliters (mL) saline as a constant rate intravenous (IV) infusion of 60 minutes.
- Cohort 1: 900 mg Linezolid: 450 mL Zyvox plus 150 mL saline as a constant rate IV infusion of 60 minutes.
- Cohort 1: 1200 mg Linezolid: 600 mL Zyvox as a constant rate IV infusion of 60 minutes.
Arm/Group | Cohort 1: Placebo | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9 | 9
participants
  AEs | 1 | 3 | 2
  SAEs | 0 | 0 | 0

2. Secondary Outcome: Cohort 1: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC Inf) and Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC Last)
Description: AUC inf = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time.
  AUC last = Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Time Frame: predose, 30 minutes, and at 1 (end of infusion), 1.5, 2, 3, 4, 6, 8, 12, 24, and 46 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: microgram (ug)*hours (hr)/mL
Arm/Group | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9
microgram (ug)*hours (hr)/mL
  AUC inf | 223.49 (47.372) | 346.89 (77.867)
  AUC last | 211.26 (48.542) | 332.26 (71.313)

3. Secondary Outcome: Cohort 1: Maximum Observed Plasma Concentration (Cmax)
Time Frame: predose, 30 minutes, and at 1 (end of infusion), 1.5, 2, 3, 4, 6, 8, 12, 24, and 46 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9
ug/mL | 22.3 (3.681) | 29.37 (6.080)

4. Secondary Outcome: Cohort 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) and Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: predose, 30 minutes, and at 1 (end of infusion), 1.5, 2, 3, 4, 6, 8, 12, 24, and 46 hours after start of infusion
Population: PK parameter analysis population
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9
hr
  Tmax | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 1.52]
  t1/2 | 6.9 [5.0 to 10.3] | 7.1 [5.1 to 11.9]

5. Secondary Outcome: Cohort 1: Clearance of Linezolid (CL)
Description: Drug clearance = Dose / AUC inf
Time Frame: predose, 30 minutes, and at 1 (end of infusion), 1.5, 2, 3, 4, 6, 8, 12, 24, and 46 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: mL/minute (min)/kilogram (kg)
Arm/Group | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9
mL/minute (min)/kilogram (kg) | 1.0173 (0.14637) | 0.8813 (0.16623)

6. Secondary Outcome: Cohort 1: Steady-State Volume of Distribution (Vss)
Description: Vss = (mean residence time [The average total time molecules of a given dose spend in the body] extrapolated to infinity) multiplied by CL
Time Frame: predose, 30 minutes, and at 1 (end of infusion), 1.5, 2, 3, 4, 6, 8, 12, 24, and 46 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid
Number analyzed (Participants) | 9 | 9
L/kg | 0.6016 (0.06869) | 0.5776 (0.04605)

7. Primary Outcome: Cohort 2: Mean Time-Matched Difference in Time Corresponding to Beginning of Depolarization to Repolarization of the Ventricles, Corrected for Heart Rate Using Fridericia's Formula (QTcF Interval) Between Linezolid 600 mg and 1200 mg Compared to Placebo
Description: The time corresponding to the beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for ventricular rate (VR) using the QT and VR from each electrocardiogram by Fridericia's formula (QTcF = QT divided by cube root of VR in seconds). A measure of dispersion is not available.
Time Frame: 0.5, 1, 2, 4, 8, 12, 24 hours post-dose
Population: The pharmacokinetic (PK) parameter analysis population was defined as all subjects randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Number; unit: milliseconds (msec)
Groups:
- Cohort 2: 600 mg Linezolid; Cohort 2: 1200 mg Linezolid: Zyvox IV Injection
- Cohort 2: Placebo: 0.9% Saline
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid | Cohort 2: Placebo
Number analyzed (Participants) | 40 | 40 | 40
milliseconds (msec)
  0.5 hour | 421.31 | 422.34 | 419.84
  1 hour | 419.71 | 420.89 | 422.67
  2 hours | 414.27 | 412.30 | 419.80
  4 hours | 418.85 | 421.92 | 418.45
  8 hours | 409.75 | 412.25 | 411.13
  12 hours | 412.99 | 413.45 | 411.98
  24 hours | 414.83 | 417.27 | 415.47
Statistical Analysis 1: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 0.5 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.47, 90% CI [-0.7 to 3.64]
Statistical Analysis 2: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 1 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -2.96, 90% CI [-5.13 to -0.79]
Statistical Analysis 3: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 2 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -5.53, 90% CI [-7.70 to -3.36]
Statistical Analysis 4: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 4 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 0.40, 90% CI [-1.77 to 2.57]
Statistical Analysis 5: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 8 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -1.37, 90% CI [-3.54 to 0.80]
Statistical Analysis 6: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 12 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.01, 90% CI [-1.16 to 3.18]
Statistical Analysis 7: Comparison: Cohort 2: 600 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 24 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -0.64, 90% CI [-2.81 to 1.53]
Statistical Analysis 8: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 0.5 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 2.49, 90% CI [0.32 to 4.66]
Statistical Analysis 9: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 1 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -1.78, 90% CI [-3.95 to 0.39]
Statistical Analysis 10: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 2 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -7.51, 90% CI [-9.68 to -5.34]
Statistical Analysis 11: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 4 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 3.47, 90% CI [1.30 to 5.64]
Statistical Analysis 12: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 8 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.13, 90% CI [-1.04 to 3.30]
Statistical Analysis 13: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 12 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.47, 90% CI [-0.70 to 3.64]
Statistical Analysis 14: Comparison: Cohort 2: 1200 mg Linezolid vs Cohort 2: Placebo; Inferential analysis at 24 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.80, 90% CI [-0.37 to 3.97]

8. Secondary Outcome: Cohort 2: Mean Time-Matched Difference in QTcF Intervals Between Moxifloxacin and Placebo
Description: A measure of dispersion is not available.
Time Frame: 0.5, 1, 2, 4, 8, 12, 24 hours post-dose
Population: PK parameter analysis population
Measure: Number; unit: msec
Groups:
- Cohort 2: Moxifloxacin: Oral administration, positive control, not blinded.
Arm/Group | Cohort 2: Moxifloxacin | Cohort 2: Placebo
Number analyzed (Participants) | 40 | 40
msec
  0.5 hour | 423.11 | 419.84
  1 hour | 429.50 | 422.67
  2 hours | 430.07 | 419.80
  4 hours | 428.29 | 418.45
  8 hours | 420.53 | 411.13
  12 hours | 419.02 | 411.98
  24 hours | 421.99 | 415.47
Statistical Analysis 1: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 0.5 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 3.27, 90% CI [1.10 to 5.44]
Statistical Analysis 2: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 1 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 6.83, 90% CI [4.66 to 9.00]
Statistical Analysis 3: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 2 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 10.27, 90% CI [8.10 to 12.44]
Statistical Analysis 4: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 4 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 9.84, 90% CI [7.67 to 12.01]
Statistical Analysis 5: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 8 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 9.40, 90% CI [7.23 to 11.58]
Statistical Analysis 6: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 12 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 7.05, 90% CI [4.87 to 9.22]
Statistical Analysis 7: Comparison: Cohort 2: Moxifloxacin vs Cohort 2: Placebo; Inferential analysis at 24 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 6.52, 90% CI [4.35 to 8.69]

9. Secondary Outcome: Cohort 2: Mean Time-Matched Difference in Uncorrected QT Intervals Between Linezolid 600 mg and 1200 mg Compared to Placebo
Description: A measure of dispersion is not available.
Time Frame: 0.5, 1, 2, 4, 8, 12, 24 hours post-dose
Population: PK parameter analysis population
Measure: Number; unit: msec
Arm/Group | Cohort 2: Placebo | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40 | 40
msec
  0.5 hour | 424.08 | 422.60 | 420.60
  1 hour | 422.25 | 414.80 | 410.06
  2 hours | 421.15 | 415.40 | 406.76
  4 hours | 420.58 | 419.66 | 418.40
  8 hours | 405.30 | 399.66 | 406.40
  12 hours | 398.85 | 396.56 | 398.96
  24 hours | 416.38 | 415.80 | 419.06
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 0.5 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -1.49, 90% CI [-5.54 to 2.57]
Statistical Analysis 2: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 1 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -7.45, 90% CI [-11.51 to -3.40]
Statistical Analysis 3: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 2 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -5.75, 90% CI [-9.81 to -1.70]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 4 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -0.92, 90% CI [-4.97 to 3.13]
Statistical Analysis 5: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 8 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -5.64, 90% CI [-9.69 to -1.58]
Statistical Analysis 6: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 12 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -2.29, 90% CI [-6.34 to 1.77]
Statistical Analysis 7: Comparison: Cohort 2: Placebo vs Cohort 2: 600 mg Linezolid; Inferential analysis at 24 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -0.59, 90% CI [-4.64 to 3.47]
Statistical Analysis 8: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 0.5 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -3.49, 90% CI [-7.54 to 0.57]
Statistical Analysis 9: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 1 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -12.19, 90% CI [-16.24 to -8.13]
Statistical Analysis 10: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 2 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -14.39, 90% CI [-18.44 to -10.33]
Statistical Analysis 11: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 4 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = -2.19, 90% CI [-6.24 to 1.87]
Statistical Analysis 12: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 8 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 1.10, 90% CI [-2.95 to 5.15]
Statistical Analysis 13: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 12 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 0.11, 90% CI [-3.94 to 4.17]
Statistical Analysis 14: Comparison: Cohort 2: Placebo vs Cohort 2: 1200 mg Linezolid; Inferential analysis at 24 hour post-dose; Test type: Superiority or Other; Mean Difference (Final Values) = 2.68, 90% CI [-1.37 to 6.73]

10. Secondary Outcome: Cohort 2: AUC Inf and AUC Last
Description: as for outcome 2
Time Frame: Predose, 30 minutes, 1, 2, 4, 8, 12 hours post-dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ug *hr/mL
Arm/Group | Cohort 2: 900 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40
ug *hr/mL
  AUC Inf | 141.75 (36.156) | 328.75 (79.198)
  AUC Last | 129.52 (32.121) | 299.40 (62.096)

11. Secondary Outcome: Cohort 2: Cmax
Time Frame: Predose, 30 minutes, 1, 2, 4, 8, 12 hours post-dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40
ug/mL | 15.06 (2.616) | 30.76 (4.395)

12. Secondary Outcome: Cohort 2: Tmax and t1/2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Tmax is the time to reach Cmax.
Time Frame: Predose, 30 minutes, 1, 2, 4, 8, 12 hours post-dose
Population: PK parameter analysis population
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40
hr
  Tmax | 1.083 [1.0 to 2.0] | 1.1 [1.0 to 2.0]
  t1/2 | 6.095 [2.83 to 10.40] | 6.796 [3.12 to 10.50]

13. Secondary Outcome: Cohort 2: CL
Description: Drug clearance = Dose / AUC inf
Time Frame: Predose, 30 minutes, 1, 2, 4, 8, 12 hours post-dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40
mL/min/kg | 1.2825 (0.36529) | 1.1000 (0.27875)

14. Secondary Outcome: Cohort 2: Vss
Description: as for outcome 6
Time Frame: Predose, 30 minutes, 1, 2, 4, 8, 12 hours post-dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid
Number analyzed (Participants) | 40 | 40
L/kg | 0.6418 (0.08353) | 0.6185 (0.06560)

15. Secondary Outcome: Cohort 2: Number of Subjects With AEs and SAEs
Description: as for outcome 1
Time Frame: From the time the subject had taken at least one dose of study treatment up to 5 weeks
Population: SAS
Measure: Number; unit: participants
Arm/Group | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid | Cohort 2: Placebo | Moxifloxacin 400 mg
Number analyzed (Participants) | 40 | 40 | 40 | 40
participants
  AEs | 3 | 7 | 4 | 10
  SAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1: Placebo | Cohort 1: 900 mg Linezolid | Cohort 1: 1200 mg Linezolid | Cohort 2: Placebo | Cohort 2: 600 mg Linezolid | Cohort 2: 1200 mg Linezolid | Cohort 2: 400 mg Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/9 | 3/9 | 2/9 | 4/40 | 3/40 | 7/40 | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=9) | Cohort 1: 900 mg Linezolid (N=9) | Cohort 1: 1200 mg Linezolid (N=9) | Cohort 2: Placebo (N=40) | Cohort 2: 600 mg Linezolid (N=40) | Cohort 2: 1200 mg Linezolid (N=40) | Cohort 2: 400 mg Moxifloxacin (N=40)
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.